CLINICAL TRIAL: NCT02043587
Title: A Phase II Study of Punctual, Cyclic, and Intensive Chemotherapy With Liposomal Cytarabine (Depocyt®) CNS Prophylaxis for Adults With Acute Lymphoblastic Leukemia and Lymphoblastic Lymphoma
Brief Title: Chemotherapy With Liposomal Cytarabine CNS Prophylaxis for Adult Acute Lymphoblastic Leukemia & Lymphoblastic Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Original investigator for the trial has left
Sponsor: University of California, San Diego (Other)
Collaborators: Leadiant Biosciences, Inc. (Industry)
Responsible Party: Principal Investigator, James Mangan, Associate Clinical Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130934
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Acute Lymphocytic Leukemia; Adult Lymphoblastic Lymphoma
Keywords: Acute lymphoblastic leukemia; Lymphoblastic leukemia; Lymphoblastic lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Daunorubicin; Vincristine; pegaspargase; Cyclophosphamide; Prednisone; Methotrexate; Leucovorin; Cytarabine; Etoposide; Dasatinib; Rituximab; Hydrocortisone; hydrocortisone hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy for ALL (Experimental): Course 1A: DNR 60 mg/m2 IV d1,2,3; VCR 1.4 mg/m2 d1,8,15,22 (cap 2 mg age >50); PEG-asp 2000 IU/m2 IV d16, age >50 1000 IU/m2, cap 3750 IU/m2; CTX 750 mg/m2 d1,15 age < 40; Prednisone 60 mg/m2 PO d1-28; Liposomal AraC 25 mg IT d1, 15
  1B: MTX 220 mg/m2 IV then 60 mg/m2/h for 36h d2-3,d16-17; LCV 50 mg/m2 IV q6h x3 then 10 mg/m2 PO/IV q6h til MTX <0.1 uM; 6-MP 60 mg/m2 PO d2-8, d16-22; PEG-asp 2000 IU/m2 IV d18, age >50 1000 IU/m2, cap 3750 IU/m2
  1C: AraC 2 g/m2 IV d1-4; Etoposide 500 mg/m2 IV d1-4
  1A-C repeat x1(2A-C) then 3rd Course B (3B)
  Maintenance (monthly, 24 mo): Prednisone 60 mg/m2 PO d1-5; VCR 1.4 mg/m2 IV d1 (cap 2 mg age >50); MTX 20 mg/m2 PO wkly; 6-MP 60 mg/m2 PO qd PEG-asp 2000 IU/m2 IV d16, age >50 1000 IU/m2, cap 3,750 IU/m2 (Mo. 1)
  Maintenance mo. 1-4: Liposomal AraC 50 mg IT d1
  Dasatinib 140 mg PO qd if Ph/BCR-ABL+; Rituximab 375 mg/m2 IV d1,15 of 1A-C, 2A (Pre-B)
  1:1 randomization: hydrocortisone v. placebo before PEG-asp 1B, 2B, & Maint.
  Interventions: Drug: DNR; Drug: VCR; Drug: PEG-asp; Drug: CTX; Drug: Prednisone; Drug: Liposomal AraC; Drug: MTX; Drug: LCV; Drug: AraC; Drug: Etoposide; Drug: Dasatinib; Drug: Rituximab; Drug: Hydrocortisone

INTERVENTIONS:
Drug: DNR — Daunorubicin 60 mg/m2 IV (in the vein) daily 1,2,3 Courses 1A, 2A
  Other Names: Daunorubicin; Daunorubicin Hydrochloride; Cerubidine; Daunomycin; Rubidomycin
Drug: VCR — 1.4 mg/m2 IV, days 1, 8, 15, 22 (cap at 2mg for ages >50) during Courses 1A, 2A; Maintenance: Day 1 during months 2-12
  Other Names: Vincristine; Oncovin; Vincasar; PFS; Vincrex; Leurocritine; LCR
Drug: PEG-asp — 2,000 IU/m2 IV for ages </= 50, age > 50, 1000 IU/m2 IV Day 16, Courses 1A & 2A; Day 18, Course 1B; Day 17, Course 2B; Day 16, Maintenance, Month 1
  Other Names: PEG-L-asparaginase; Oncaspar; PEG-asparaginase; pegasparagase
Drug: CTX — 750 mg/m2 IV, days 1 &15 for subjects <40 year of age, substitute cyclophosphamide 500 mg/m2 IV over 60 minutes every 12 hours for 4 doses on days 15 & 16 for subjects < 40 years of age if day 14 bone marrow M2 or M3; Courses 1A & 2A
  Other Names: Cyclophosphamide; Cytoxan; Endoxan; Neosar; Procytox; Revimmune; cytophosphane; CPM; CYT
Drug: Prednisone — 60 mg/m2 orally once daily on days 1-28 during Courses 1A & 2A; Maintenance: Monthly, days 1-5
  Other Names: Deltasone
Drug: Liposomal AraC — 25 mg intrathecal (IT), on days 1 & 15 during Courses 1A & 2A; 50 mg intrathecal on day 1 during Maintenance Months 1 through 4
  Other Names: Liposomal cytarabine; DepoCyt
Drug: MTX — 220 mg/m2 IV bolus over 15 minutes then 60 mg/m2/hour for 36 hours once on days 2-3 and 16-17 during Courses 1B & 2B; 20 mg/m2 orally one day per week every 7 days during Maintenance Months
  Other Names: Methotrexate; Rheumatrex; Trexall
Drug: LCV — 50 mg/m2 IV over 15-30 minutes every 6 hours for 3 doses to begin immediately after completion of methotrexate infusion, then 10 mg/m2 orally or IV over 15-30 minutes every 6 hours until methotrexate level less than 0.1 micromolar during Courses 1B & 2B
  Other Names: Leucovorin
Drug: AraC — 2,000 mg/m2 IV, days 1-4 during Courses 1C & 2C
  Other Names: Cytarabine; Ara-C; Arabinosylcytosine; Cytosar-U
Drug: Etoposide — 500 mg/m2 IV over 3 hours once daily on days 1-4 during Courses 1C & 2C
  Other Names: VP-16; VePesid; Toposar
Drug: Dasatinib — 140 mg orally daily if BCR/ABL positive and/or Ph+
  Other Names: Sprycel
Drug: Rituximab — 375 mg/m2 IV once daily on days 1 & 15 (precursor B-cell ALL only, administer per institutional protocol) during Courses 1A, 1B, 1C & 2A
  Other Names: Rituxan
Drug: Hydrocortisone — Randomize patients proceeding to Course 1B to hydrocortisone versus placebo prior to PEG-asparaginase treatments in Courses 1B, 2B, 3B, and Maintenance month 1
  Other Names: Hydrocortisone sodium succinate; Solu-Cortef

SUMMARY:
The objective of this protocol is to improve survival for adults with acute lymphoblastic leukemia or acute lymphoblastic lymphoma by reducing systemic and central nervous system (CNS) relapse with acceptable toxicity using intensive chemotherapy with liposomal cytarabine (Depocyt®) CNS prophylaxis.

DETAILED DESCRIPTION:
This treatment regimen builds on the "Linker" regimen/UCSF Protocol 8707 ALL regimen backbone with the goal of improved efficacy and acceptable toxicity by substituting pegylated asparaginase for native L-asparaginase, the addition of rituximab for pre-B-cell ALL, and the addition of dasatinib for Philadelphia chromosome/BCR-ABL positive ALL, and the addition of cyclophosphamide for younger adults. In addition, the study regimen aims to reduce CNS relapse through the use of intrathecal liposomal cytarabine in place of intrathecal methotrexate for CNS relapse prophylaxis and

The regimen uses 3 modules of therapy with non-cross-resistant chemotherapy agents. Rituximab is added for a total of 8 doses for patients with pre-B-cell ALL. Dasatinib is added for patients with Ph+ ALL.

Course 1A (Induction): Daunorubicin, vincristine, PEG-asparaginase, and prednisone for all patients with the addition of cyclophosphamide for patients 18-39 years of age. Treatment is intensified for patients with disease present on a day 14 bone marrow biopsies during Induction Course 1A. In addition to standard analyses, minimal residual disease will be assessed on day 14 and remission bone marrow aspirates and correlated with outcomes.

Course 1B: High-dose methotrexate, oral 6-mercaptopurine, and PEG-asparaginase.

Course 1C: High-dose cytarabine and etoposide.

The 3 courses then repeat (2A (Intensification), 2B, 2C) followed by a final "B" cycle (3B) of high-dose methotrexate, 6-mercaptopurine, and PEG-asparaginase.

After completion of Course 3B, patients proceed to maintenance chemotherapy with monthly methotrexate, vincristine, 6-mercaptopurine, and prednisone cycles for 24 months with a single dose PEG-asparaginase given in month 1 of Maintenance.

CNS prophylaxis: Intrathecal liposomal cytarabine replaces intrathecal methotrexate CNS prophylaxis and is given every 2 weeks during the "A" Induction and Intensification courses then every 3 months during Maintenance for a total of 8 doses. Given the presence of CNS penetrating chemotherapy in the "B" and "C" cycles, intrathecal liposomal cytarabine is not given due to risk of excessive CNS toxicity.

There is a randomization to hydrocortisone or placebo premedication prior to PEG-asparaginase.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent.
* Diagnosis of acute lymphoblastic leukemia or lymphoblastic lymphoma as defined by the World Health Organization [94]
* Untreated disease EXCEPT for corticosteroids, hydroxyurea, leukapheresis, and/or tyrosine kinase inhibitors for up to 2 weeks prior to initiation of study therapy.
* Age 18 through 60 years
* ECOG performance status 0,1, or 2 (see Appendix A)
* Adequate organ function defined as:
* Total bilirubin < 2 mg/dL (unless due to ALL)
* AST(SGOT)/ALT(SGPT) < 3 times institutional upper limit of normal (unless due to ALL)
* Serum creatinine < 2 mg/dL (unless elevated creatinine felt by investigator to be acute and reversible) OR creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Left ventricular ejection fraction ≥50%
* Women of child-bearing potential and men with partners of child- bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)

Exclusion Criteria:

* Current or anticipated use of other investigational agents during the study
* Known central nervous system mass lesion
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to liposomal cytarabine or other agents used in study inclusive of known allergy to polyethylene glycol.
* History of unprovoked venous thrombosis/thromboembolism
* Recurrent or chronic pancreatitis
* Uncontrolled diabetes mellitus
* Uncontrolled intercurrent illness that would limit compliance with study requirements including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing.
* Any condition, in the opinion of the investigator, that compromises compliance with study requirements
* Known HIV positivity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-01; Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 3-year

SECONDARY OUTCOMES:
Liposomal cytarabine toxicity | 3 years
CNS relapse rate | 3-year
Overall survival | 3-year
Leukemia-free survival | 3-year
Efficacy of hydrocortisone premedication for reduced PEG-asparaginase allergic reactions | 3 years
PEG-asparaginase toxicities | 3 years
Complete and overall response rates | 3 years
Non-relapse mortality | 3-year

OTHER OUTCOMES:
Minimal residual disease and outcomes | 3 years
Asparaginase antibodies and asparaginase activity | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: James K Mangan, MD, PhD, Principal Investigator — UC San Diego, Division of Blood and Marrow Transplantation
Locations (4):
- United States (4):
  - UCSD, Division of Blood and Marrow Transplantation, Moores Cancer Center, La Jolla, California
  - Hematological Malignancies/Stem Cell Transplantation Unit, David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Comprehensive Cancer Center, San Francisco, California

REFERENCES:
- [Result] Linker C, Damon L, Ries C, Navarro W. Intensified and shortened cyclical chemotherapy for adult acute lymphoblastic leukemia. J Clin Oncol. 2002 May 15;20(10):2464-71. doi: 10.1200/JCO.2002.07.116. PMID 12011123